CLINICAL TRIAL: NCT00002143
Title: Treatment of Psoriasis Using Acitretin in HIV-Positive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 239A; 65-93(2)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: HIV Infections; Psoriasis
Keywords: Psoriasis; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Acitretin
MeSH Terms: conditions — HIV Infections; Psoriasis; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Acitretin

INTERVENTIONS:
Drug: Acitretin

SUMMARY:
To determine the efficacy of acitretin in the treatment of psoriasis in HIV/AIDS patients.

Etretinate, a retinoid, has proven successful in the treatment of HIV-infected patients with psoriasis, but it has an elimination half-life of 100 days. Acitretin, a metabolite of etretinate, has a much shorter half-life of 2 to 3 days. Acitretin has proven effective in treating psoriasis in patients without HIV infection by reducing skin involvement and clearing of the condition, but it has not been thoroughly evaluated in HIV-infected patients.

DETAILED DESCRIPTION:
Etretinate, a retinoid, has proven successful in the treatment of HIV-infected patients with psoriasis, but it has an elimination half-life of 100 days. Acitretin, a metabolite of etretinate, has a much shorter half-life of 2 to 3 days. Acitretin has proven effective in treating psoriasis in patients without HIV infection by reducing skin involvement and clearing of the condition, but it has not been thoroughly evaluated in HIV-infected patients.

Patients receive acitretin daily, with dose increases every 4 weeks based on quantitative assessment of the skin using the Psoriasis Area and Severity Index (PASI). Treatment continues for a total of 20 weeks. Patients are followed every 2 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Any nondermatologic medication.

Patients must have:

* HIV infection.
* Psoriasis involving at least 10 percent of body surface.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Med Ctr, New York, New York, United States